CLINICAL TRIAL: NCT01335958
Title: A Phase I, Open-Label, Dose Escalation Study of the Safety and Pharmacokinetics of DMUC5754A Administered Intravenously to Patients With Platinum-Resistant Ovarian Cancer or Unresectable Pancreatic Cancer
Brief Title: Safety and Pharmacokinetics of DMUC5754A Administered Intravenously to Patients With Platinum-Resistant Ovarian Cancer or Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DGR4980g; GO00766 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Ovarian Cancer, Pancreatic Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Pancreatic Neoplasms | interventions — DMUC5754A

ARMS (1):
- A (Experimental)
  Interventions: Drug: DMUC5754A

INTERVENTIONS:
Drug: DMUC5754A — Escalating intravenous dose

SUMMARY:
This is a Phase I, multi-center, open-label, dose-escalation study of DMUC5754A administered as a single agent by intravenous (IV) infusion to patients with platinum-resistant ovarian cancer or unresectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Documented willingness to use an effective means of contraception for women of childbearing potential
* Measurable disease with at least one lesion that can be accurately measured in at least one dimension

Inclusion Criteria Specific to Patients with Ovarian Cancer:

* Advanced, epithelial ovarian, primary peritoneal, or fallopian tube cancer that has progressed or relapsed during or within 6 months of the most recent treatment with a platinum-containing chemotherapy regimen, and for which no standard therapy exists
* For patients in the dose-expansion cohort of the study only, no more than two prior chemotherapy regimens for the treatment of platinum-resistant ovarian cancer

Inclusion Criteria Specific to Patients with Pancreatic Cancer:

* Incurable, locally advanced, or metastatic disease for which no standard therapy exists, consisting of unresectable pancreatic ductal adenocarcinoma, including recurrence of previously-resected disease that is considered unresectable with curative intent
* No more than one chemotherapy regimen (approved or experimental) administered in the metastatic setting

Exclusion Criteria:

* Anti-tumor therapy, including chemotherapy, biologic, experimental, or hormonal therapy within 4 weeks prior to Day 1
* Palliative radiation to bone metastases within 2 weeks prior to Day 1
* Major surgical procedure within 4 weeks prior to Day 1
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including HIV and atypical mycobacterial disease, but excluding fungal infections of the nail beds)
* Current Grade >1 toxicity (except alopecia and anorexia) from prior therapy or Grade >1 neuropathy from any cause
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided that they meet all of the following criteria: evaluable or measurable disease outside the CNS, radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study, and the screening CNS radiographic study is >= 8 weeks since completion of radiotherapy and >= 4 weeks since the discontinuation of corticosteroids and anticonvulsants.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Evidence of significant uncontrolled concomitant diseases, such as cardiovascular disease (including stroke, New York Heart Association Class III or IV cardiac disease or myocardial infarction within 6 months prior to screening, unstable arrhythmias, and unstable angina); nervous system, pulmonary (including obstructive pulmonary disease and history of symptomatic bronchospasm), renal, hepatic, endocrine, or gastrointestinal disorders; or a serious non-healing wound or fracture
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to 21 days
Nature of dose-limiting toxicities (DLTs) graded per NCI CTCAE v4.0 | Up to 21 days

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 1 year
Nature of adverse events graded per NCI CTCAE v4.0 | Up to 1 year
Severity of adverse events | Up to 1 year
Area under the concentration-time curve | up to 1 year
Maximum concentrations | up to 1 year
Minimum concentrations | up yo 1 year
Clearance | up to 1 year
Half-life | up to 1 year
Volume of distribution | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (3):
- United States (3):
  - Boston, Massachusetts
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee

REFERENCES:
- [Derived] Liu JF, Moore KN, Birrer MJ, Berlin S, Matulonis UA, Infante JR, Wolpin B, Poon KA, Firestein R, Xu J, Kahn R, Wang Y, Wood K, Darbonne WC, Lackner MR, Kelley SK, Lu X, Choi YJ, Maslyar D, Humke EW, Burris HA. Phase I study of safety and pharmacokinetics of the anti-MUC16 antibody-drug conjugate DMUC5754A in patients with platinum-resistant ovarian cancer or unresectable pancreatic cancer. Ann Oncol. 2016 Nov;27(11):2124-2130. doi: 10.1093/annonc/mdw401. PMID 27793850